CLINICAL TRIAL: NCT04382326
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY INFANTS
Brief Title: 20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study of a 4-Dose Series in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B7471011; 2019-003305-10 (EudraCT Number)
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20-valent pneumococcal conjugate vaccine (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine
- 13-valent pneumococcal conjugate vaccine (Active Comparator): Pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — 20-valent pneumococcal conjugate vaccine
  Arms: 20-valent pneumococcal conjugate vaccine
Biological: 13-valent pneumococcal conjugate vaccine — 13-valent pneumococcal conjugate vaccine
  Arms: 13-valent pneumococcal conjugate vaccine

SUMMARY:
20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study of a 4-Dose Series in Healthy Infants

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at >36 weeks of gestation and 2 months of age at the time of consent.
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis)
* Major known congenital malformation or serious chronic disorder
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results
* Previous receipt of >1 dose of hepatitis B vaccine; or receipt of a single hepatitis B vaccine dose administered at >30 days old, or previous receipt of any licensed or investigational pneumococcal vaccine, or planned receipt through study participation

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1997 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (108):
- United States (103):
  - Children's of Alabama, Birmingham, Alabama
  - UAB Pediatric Primary Care Clinic at Children's of Alabama, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - MedPharmics, LLC, Phoenix, Arizona
  - Northwest Arkansas Pediatrics, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Gardens Medical Center, Bell Gardens, California
  - Coast Clinical Research, LLC, Bellflower, California
  - Priti Desai, M.D. Inc., Covina, California
  - Universal Biopharma Research Institute Inc., Fresno, California
  - Matrix Clinical Research, Gardena, California
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Kaiser Permanente Oakland, Oakland, California
  - Orange County Research Institute, Ontario, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Children's Colorado Health Pavilion (Child Health Clinic), Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - Optumcare Colorado Springs, LLC, Colorado Springs, Colorado
  - Gentle Medicine Associates, Boynton Beach, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Benton Pediatrics, Gainesville, Florida
  - Qway Research, Hialeah, Florida
  - Next Phase Research Alliance, Homestead, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Crystal Biomedical Research, LLC, Miami Lakes, Florida
  - Children's Health Center, Tampa, Florida
  - Tekton Research, Inc, Chamblee, Georgia
  - Uptown Pediatrics, Columbus, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Meridian Clinical Research, Macon, Georgia
  - Omega Pediatrics, Roswell, Georgia
  - Idaho Falls Pediatrics, Ammon, Idaho
  - Idaho Falls Pediatrics, Idaho Falls, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Family First Medical Center, Idaho Falls, Idaho
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - The Pediatric Center, Idaho Falls, Idaho
  - Saltzer Health, Nampa, Idaho
  - ASR, LLC, Nampa, Idaho
  - The Iowa Clinic, Ankeny, Iowa
  - Blank Children's Pediatric Clinic, Des Moines, Iowa
  - Unity Point Health, Des Moines, Iowa
  - The Iowa Clinic, West Des Moines, Iowa
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Michael W. Simon, MD, PSC, Lexington, Kentucky
  - Novak Center for Children's Health, Louisville, Kentucky
  - Brownsboro Park Pediatrics, Louisville, Kentucky
  - Velocity Clinical Research at Primary Pediatrics, Macon, Baton Rouge, Louisiana
  - Benchmark Research, Covington, Louisiana
  - ACC Pediatric Research, Haughton, Louisiana
  - Velocity Clinical Research, Covington, Metairie, Louisiana
  - University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - The Pediatric Center of Frederick, LLC, Frederick, Maryland
  - MedPharmics, LLC, Gulfport, Mississippi
  - Boeson Research, Missoula, Montana
  - Meridian Clinical Research, Hastings, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Children's Physicians Dundee, Omaha, Nebraska
  - Medpharmics, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Child Health Care Associates, East Syracuse, New York
  - Smart Medical Research, Inc, Jackson Heights, New York
  - Child Health Care Associates, Liverpool, New York
  - ECU Physicians Adult and Pediatric Health Center, Greenville, North Carolina
  - ECU Physicians Pediatric Outpatient Clinic, Greenville, North Carolina
  - Leo Jenkins Cancer Center Pharmacy, Greenville, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association, Inc., Dayton, Ohio
  - Pediatric Associates of Fairfield, Fairfield, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Pediatric Medical Associates, East Norriton, Pennsylvania
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Lockman & Lubell Pediatric Associates, Fort Washington, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Palmetto Pediatrics, PA, North Charleston, South Carolina
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - Sanford 69th & Louise Family Medicine, Sioux Falls, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - Premier Medical Group, Clarksville, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Coastal Bend Clinical Research, Corpus Christi, Texas
  - Kool Kids Pediatrics, Houston, Texas
  - La Providence Pediatrics Clinic, Houston, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Diagnostic Clinic of Longview, Longview, Texas
  - Ashley Pediatrics Day and Night Clinic, McAllen, Texas
  - Dr. Ruben Aleman & Associates, McAllen, Texas
  - Tekton Research, Inc, San Antonio, Texas
  - Wee Care Pediatrics, Kaysville, Utah
  - Wee Care Pediatrics, Layton, Utah
  - Wasatch Pediatrics, Cottonwood Office, Murray, Utah
  - Wee Care Pediatrics, Roy, Utah
  - Dixie Pediatrics, St. George, Utah
  - Wee Care Pediatrics, Syracuse, Utah
  - Pediatric Associates of Charlottesville, PLC, Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - The Vancouver Clinic, Inc, Vancouver, Washington
- Puerto Rico (5):
  - San Miguel Medical, Trujillo Alto, PR
  - Cooperativa de Facultad Medica Sanacoop DBA Instituto Sanacoop, Bayamón
  - Clinical Research Puerto Rico, Guayama
  - Hispanic Alliance for Clinical and Translational Research, San Juan
  - San Juan Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Senders S, Korbal P, Kline M, Tamimi N, Thompson A, Drozd J, Cutler MW, Giardina PC, Trammel J, Lei L, Peng Y, Watson W, McElwee K. Immunogenicity and safety of concomitant vaccines given with 20-valent pneumococcal conjugate vaccine in healthy infants. Vaccine. 2025 Dec 5;68:127916. doi: 10.1016/j.vaccine.2025.127916. Epub 2025 Nov 3. PMID 41187484
- [Derived] Senders S, Klein NP, Tamimi N, Thompson A, Baugher G, Trammel J, Peng Y, Giardina P, Scully IL, Pride M, Center KJ, Gruber WC, Scott DA, Watson W. A Phase Three Study of the Safety and Immunogenicity of a Four-dose Series of 20-Valent Pneumococcal Conjugate Vaccine in Healthy Infants. Pediatr Infect Dis J. 2024 Jun 1;43(6):596-603. doi: 10.1097/INF.0000000000004334. Epub 2024 Mar 26. PMID 38535409
- [Derived] Mt-Isa S, Chumbley JR, Crawford EL, Banniettis N, Buchwald UK, Weaver J, Weiss T. An indirect treatment comparison (ITC) and matching-adjusted indirect comparison (MAIC) between a 15-valent (V114) and a 20-valent (PCV20) pneumococcal conjugate vaccine among healthy infants. Expert Rev Vaccines. 2023 Jan-Dec;22(1):906-917. doi: 10.1080/14760584.2023.2270039. Epub 2023 Oct 19. PMID 37846456
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1997 participants were enrolled and assigned to receive 4 doses of 20-valent pneumococcal conjugate vaccine (20vPnC) or 13vPnC of which 6 participants were not vaccinated and 1991 were vaccinated with either 20vPnC or 13vPnC.
Groups:
- 20vPnC: Infants 42 to 98 days of age were enrolled to receive 4 doses of 0.5 millilitre (mL) 20-valent Pneumococcal Conjugate Vaccine (20vPnC) intramuscularly. Dose 1 was given at enrollment and Dose 2 and 3 were given 42 to 63 days from the previous dose. Dose 4 was administered at 365 to 455 days of age.
- 13vPnC: Infants 42 to 98 days of age were enrolled to receive 4 doses of 0.5 millilitre (mL) 13-valent Pneumococcal Conjugate Vaccine (13vPnC) intramuscularly. Dose 1 was given at enrollment and Dose 2 and 3 were given 42 to 63 days from the previous dose. Dose 4 was administered at 365 to 455 days of age.
Period: Overall Study
Arm/Group | 20vPnC | 13vPnC
Started | 1001 | 987
Completed | 821 | 799
Not Completed | 180 | 188
Not completed — Adverse Event, not serious | 1 | 2
Not completed — Other | 1 | 0
Not completed — Withdrawal By Parent/Guardian | 50 | 54
Not completed — No Longer Meets Eligibility Criteria | 50 | 44
Not completed — Protocol Violation | 29 | 23
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 48 | 63
Not completed — Adverse Event, non-fatal | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of 20vPnC or 13vPnC and had safety data assessed after any dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20vPnC | 13vPnC | Total
Number analyzed (Participants) | 1001 | 987 | 1988
Age, Continuous [Mean (Standard Deviation); unit: Days] | 65.9 (7.98) | 65.6 (7.12) | 65.8 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 483 | 482 | 965
  Male | 518 | 505 | 1023
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 312 | 293 | 605
  Not Hispanic or Latino | 661 | 659 | 1320
  Unknown or Not Reported | 28 | 35 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 16 | 16 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 110 | 108 | 218
  White | 754 | 742 | 1496
  More than one race | 68 | 73 | 141
  Unknown or Not Reported | 47 | 43 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1
Description: Local reactions were recorded using an electronic diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were graded as mild (0.5 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement).
Time Frame: Within 7 days after Dose 1
Population: Safety population included all the participants who received at least 1 dose of the investigational product (IP) with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any electronic diary (e-diary) data reported after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 993 | 974
Percentage of participants
  Redness: Any | 25.5 [22.8 to 28.3] | 24.6 [22.0 to 27.5]
  Redness: Mild | 21.5 [18.9 to 24.1] | 22.3 [19.7 to 25.0]
  Redness: Moderate | 4.0 [2.9 to 5.4] | 2.4 [1.5 to 3.5]
  Redness: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]
  Swelling: Any | 16.4 [14.2 to 18.9] | 18.8 [16.4 to 21.4]
  Swelling: Mild | 11.5 [9.6 to 13.6] | 14.7 [12.5 to 17.1]
  Swelling: Moderate | 4.8 [3.6 to 6.4] | 4.1 [2.9 to 5.6]
  Swelling: Severe | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4]
  Pain at the injection site: Any | 49.1 [46.0 to 52.3] | 45.3 [42.1 to 48.5]
  Pain at the injection site: Mild | 30.6 [27.8 to 33.6] | 30.4 [27.5 to 33.4]
  Pain at the injection site: Moderate | 18.4 [16.1 to 21.0] | 14.9 [12.7 to 17.3]
  Pain at the injection site: Severe | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4]

2. Primary Outcome: Percentage of Participants With Local Reaction Within 7 Days After Dose 2
Description: as for outcome 1
Time Frame: Within 7 Days After Dose 2
Population: Safety population included all the participants who received at least 1 dose of the investigational product (IP) with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any electronic diary (e-diary) data reported after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 940 | 924
Percentage of participants
  Redness: Any | 23.2 [20.5 to 26.0] | 26.4 [23.6 to 29.4]
  Redness: Mild | 21.2 [18.6 to 23.9] | 23.1 [20.4 to 25.9]
  Redness: Moderate | 2.0 [1.2 to 3.1] | 3.4 [2.3 to 4.7]
  Redness: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]
  Swelling: Any | 15.5 [13.3 to 18.0] | 17.3 [14.9 to 19.9]
  Swelling: Mild | 11.5 [9.5 to 13.7] | 13.5 [11.4 to 15.9]
  Swelling: Moderate | 4.0 [2.9 to 5.5] | 3.8 [2.7 to 5.2]
  Swelling: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]
  Pain at the injection site: Any | 44.0 [40.8 to 47.3] | 41.7 [38.5 to 44.9]
  Pain at the injection site: Mild | 29.3 [26.4 to 32.3] | 27.7 [24.8 to 30.7]
  Pain at the injection site: Moderate | 14.8 [12.6 to 17.2] | 14.0 [11.8 to 16.4]
  Pain at the injection site: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3
Description: as for outcome 1
Time Frame: Within 7 days after Dose 3
Population: Safety population included all the participants who received at least 1 dose of the investigational product (IP) with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any electronic diary (e-diary) data reported after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 914 | 901
Percentage of participants
  Redness: Any | 25.4 [22.6 to 28.3] | 27.2 [24.3 to 30.2]
  Redness: Mild | 21.1 [18.5 to 23.9] | 23.5 [20.8 to 26.4]
  Redness: Moderate | 4.3 [3.1 to 5.8] | 3.7 [2.5 to 5.1]
  Redness: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]
  Swelling: Any | 17.1 [14.7 to 19.7] | 17.6 [15.2 to 20.3]
  Swelling: Mild | 12.5 [10.4 to 14.8] | 13.8 [11.6 to 16.2]
  Swelling: Moderate | 4.6 [3.3 to 6.2] | 3.8 [2.6 to 5.2]
  Swelling: Severe | 0 [0.0 to 0.4] | 0.1 [0.0 to 0.6]
  Pain at the injection site: Any | 38.6 [35.5 to 41.9] | 39.0 [35.8 to 42.2]
  Pain at the injection site: Mild | 25.7 [22.9 to 28.7] | 25.5 [22.7 to 28.5]
  Pain at the injection site: Moderate | 12.9 [10.8 to 15.3] | 13.4 [11.3 to 15.8]
  Pain at the injection site: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 4
Description: Local reactions were recorded using an electronic diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were graded as mild (0.5 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7.0 cm). Pain at injection site was graded as mild (hurt if gently touched example, whimpered, winced, protested, or withdrew), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement). 95 percent (%) confidence interval (CI) was based on Clopper and Pearson method.
Time Frame: Within 7 days after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the investigational product (IP) with safety follow up after any dose. Here, 'Number of Participants Analyzed' = number of participants with any electronic diary (e-diary) data reported after Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 826 | 815
Percentage of participants
  Redness: Any | 23.5 [20.6 to 26.5] | 26.6 [23.6 to 29.8]
  Redness: Mild | 19.6 [17.0 to 22.5] | 22.0 [19.2 to 25.0]
  Redness: Moderate | 3.9 [2.7 to 5.4] | 4.7 [3.3 to 6.3]
  Redness: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.5]
  Swelling: Any | 14.9 [12.5 to 17.5] | 17.3 [14.8 to 20.1]
  Swelling: Mild | 10.7 [8.6 to 13.0] | 13.6 [11.3 to 16.2]
  Swelling: Moderate | 4.2 [3.0 to 5.8] | 3.7 [2.5 to 5.2]
  Swelling: Severe | 0 [0.0 to 0.4] | 0 [0.0 to 0.5]
  Pain at the injection site: Any | 35.7 [32.4 to 39.1] | 35.8 [32.5 to 39.2]
  Pain at the injection site: Mild | 24.1 [21.2 to 27.2] | 27.1 [24.1 to 30.3]
  Pain at the injection site: Moderate | 11.3 [9.2 to 13.6] | 8.7 [6.9 to 10.9]
  Pain at the injection site: Severe | 0.4 [0.1 to 1.1] | 0 [0.0 to 0.5]

5. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1
Description: Systemic events included fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participant's using an e-diary. Fever was defined as temperature greater than or equal to (>=) 38.0 degrees Celsius (C) and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after Dose 1
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any e-diary data reported after Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 993 | 974
Percentage of participants
  Fever: >=38.0 degree C | 10.3 [8.5 to 12.3] | 7.5 [5.9 to 9.3]
  Fever: >=38.0 degree C to 38.4 degree C | 7.3 [5.7 to 9.0] | 6.3 [4.8 to 8.0]
  Fever: >38.4 degree C to 38.9 degree C | 2.2 [1.4 to 3.3] | 0.9 [0.4 to 1.7]
  Fever: >38.9 degree C to 40.0 degree C | 0.7 [0.3 to 1.4] | 0.3 [0.1 to 0.9]
  Fever: >40.0 degree C | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4]
  Decreased appetite: Any | 24.4 [21.7 to 27.2] | 23.9 [21.3 to 26.7]
  Decreased appetite: Mild | 14.5 [12.4 to 16.8] | 16.1 [13.9 to 18.6]
  Decreased appetite: Moderate | 9.7 [7.9 to 11.7] | 7.5 [5.9 to 9.3]
  Decreased appetite: Severe | 0.2 [0.0 to 0.7] | 0.3 [0.1 to 0.9]
  Drowsiness: Any | 67.2 [64.2 to 70.1] | 66.0 [62.9 to 69.0]
  Drowsiness: Mild | 50.2 [47.0 to 53.3] | 49.3 [46.1 to 52.5]
  Drowsiness: Moderate | 16.1 [13.9 to 18.5] | 15.6 [13.4 to 18.0]
  Drowsiness: Severe | 0.9 [0.4 to 1.7] | 1.1 [0.6 to 2.0]
  Irritability: Any | 70.9 [68.0 to 73.7] | 71.7 [68.7 to 74.5]
  Irritability: Mild | 23.4 [20.8 to 26.1] | 21.6 [19.0 to 24.3]
  Irritability: Moderate | 43.0 [39.9 to 46.1] | 46.2 [43.0 to 49.4]
  Irritability: Severe | 4.5 [3.3 to 6.0] | 3.9 [2.8 to 5.3]
  Use of antipyretic or pain medication | 35.1 [32.2 to 38.2] | 33.8 [30.8 to 36.8]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: Systemic events included fever, decreased appetite, drowsiness/increased sleep and irritability, recorded by parents/legal guardians of participant's using an e-diary. Fever was defined as temperature >= 38.0 degrees C and categorized as >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability was graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted). 95% CI was based on Clopper and Pearson method.
Time Frame: Within 7 days after Dose 2
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any e-diary data reported after Dose 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 940 | 924
Percentage of participants
  Fever: >=38.0 degree C | 17.3 [15.0 to 19.9] | 16.3 [14.0 to 18.9]
  Fever: >=38.0 degree C to 38.4 degree C | 10.9 [8.9 to 13.0] | 10.0 [8.1 to 12.1]
  Fever: >38.4 degree C to 38.9 degree C | 4.0 [2.9 to 5.5] | 4.2 [3.0 to 5.7]
  Fever: >38.9 degree C to 40.0 degree C | 2.2 [1.4 to 3.4] | 2.2 [1.3 to 3.3]
  Fever: >40.0 degree C | 0.2 [0.0 to 0.8] | 0 [0.0 to 0.4]
  Decreased appetite: Any | 26.4 [23.6 to 29.3] | 23.5 [20.8 to 26.4]
  Decreased appetite: Mild | 16.4 [14.1 to 18.9] | 15.3 [13.0 to 17.7]
  Decreased appetite: Moderate | 9.8 [8.0 to 11.9] | 7.7 [6.0 to 9.6]
  Decreased appetite: Severe | 0.2 [0.0 to 0.8] | 0.5 [0.2 to 1.3]
  Drowsiness: Any | 54.7 [51.4 to 57.9] | 55.6 [52.4 to 58.9]
  Drowsiness: Mild | 37.0 [33.9 to 40.2] | 36.9 [33.8 to 40.1]
  Drowsiness: Moderate | 16.9 [14.6 to 19.5] | 17.9 [15.4 to 20.5]
  Drowsiness: Severe | 0.7 [0.3 to 1.5] | 0.9 [0.4 to 1.7]
  Irritability: Any | 71.6 [68.6 to 74.5] | 68.8 [65.7 to 71.8]
  Irritability: Mild | 22.9 [20.2 to 25.7] | 21.2 [18.6 to 24.0]
  Irritability: Moderate | 44.7 [41.5 to 47.9] | 43.4 [40.2 to 46.7]
  Irritability: Severe | 4.0 [2.9 to 5.5] | 4.2 [3.0 to 5.7]
  Use of antipyretic or pain medication | 40.7 [37.6 to 44.0] | 41.0 [37.8 to 44.3]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3
Description: as for outcome 6
Time Frame: Within 7 days after Dose 3
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any e-diary data reported after Dose 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 914 | 901
Percentage of participants
  Fever: >=38.0 degree C | 12.6 [10.5 to 14.9] | 13.7 [11.5 to 16.1]
  Fever: >=38.0 degree C to 38.4 degree C | 7.7 [6.0 to 9.6] | 7.9 [6.2 to 9.8]
  Fever: >38.4 degree C to 38.9 degree C | 3.4 [2.3 to 4.8] | 3.9 [2.7 to 5.4]
  Fever: >38.9 degree C to 40.0 degree C | 1.4 [0.8 to 2.4] | 1.9 [1.1 to 3.0]
  Fever: >40.0 degree C | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4]
  Decreased appetite: Any | 20.6 [18.0 to 23.3] | 22.4 [19.7 to 25.3]
  Decreased appetite: Mild | 13.5 [11.3 to 15.8] | 13.9 [11.7 to 16.3]
  Decreased appetite: Moderate | 6.7 [5.1 to 8.5] | 8.2 [6.5 to 10.2]
  Decreased appetite: Severe | 0.4 [0.1 to 1.1] | 0.3 [0.1 to 1.0]
  Drowsiness: Any | 44.1 [40.8 to 47.4] | 44.1 [40.8 to 47.4]
  Drowsiness: Mild | 31.1 [28.1 to 34.2] | 30.1 [27.1 to 33.2]
  Drowsiness: Moderate | 12.5 [10.4 to 14.8] | 13.1 [11.0 to 15.5]
  Drowsiness: Severe | 0.5 [0.2 to 1.3] | 0.9 [0.4 to 1.7]
  Irritability: Any | 64.4 [61.2 to 67.5] | 63.0 [59.8 to 66.2]
  Irritability: Mild | 25.2 [22.4 to 28.1] | 21.6 [19.0 to 24.5]
  Irritability: Moderate | 37.5 [34.4 to 40.8] | 39.2 [36.0 to 42.5]
  Irritability: Severe | 1.8 [1.0 to 2.8] | 2.2 [1.4 to 3.4]
  Use of antipyretic/pain medication | 36.3 [33.2 to 39.5] | 36.1 [32.9 to 39.3]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 4
Description: as for outcome 6
Time Frame: Within 7 days after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. 'Number of Participants Analyzed' = number of participants with any e-diary data reported after Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 826 | 815
Percentage of participants
  Fever: >= 38.0 degree C | 14.5 [12.2 to 17.1] | 14.0 [11.7 to 16.6]
  Fever: >=38.0 degree C to 38.4 degree C | 6.5 [4.9 to 8.4] | 7.7 [6.0 to 9.8]
  Fever: >38.4 degree C to 38.9 degree C | 5.1 [3.7 to 6.8] | 3.2 [2.1 to 4.6]
  Fever: >38.9 degree C to 40.0 degree C | 2.7 [1.7 to 4.0] | 2.9 [1.9 to 4.4]
  Fever: >40.0 degree C | 0.2 [0.0 to 0.9] | 0.1 [0.0 to 0.7]
  Decreased appetite: Any | 24.8 [21.9 to 27.9] | 25.2 [22.2 to 28.3]
  Decreased appetite: Mild | 15.9 [13.4 to 18.5] | 16.1 [13.6 to 18.8]
  Decreased appetite: Moderate | 8.6 [6.8 to 10.7] | 8.3 [6.5 to 10.5]
  Decreased appetite: Severe | 0.4 [0.1 to 1.1] | 0.7 [0.3 to 1.6]
  Drowsiness: Any | 39.5 [36.1 to 42.9] | 39.5 [36.1 to 43.0]
  Drowsiness: Mild | 27.8 [24.8 to 31.0] | 28.2 [25.2 to 31.4]
  Drowsiness: Moderate | 11.0 [9.0 to 13.4] | 10.7 [8.6 to 13.0]
  Drowsiness: Severe | 0.6 [0.2 to 1.4] | 0.6 [0.2 to 1.4]
  Irritability: Any | 61.0 [57.6 to 64.4] | 61.1 [57.7 to 64.5]
  Irritability: Mild | 23.4 [20.5 to 26.4] | 21.8 [19.0 to 24.8]
  Irritability: Moderate | 35.0 [31.7 to 38.3] | 37.9 [34.6 to 41.3]
  Irritability: Severe | 2.7 [1.7 to 4.0] | 1.3 [0.7 to 2.4]
  Use of antipyretic/pain medication | 37.5 [34.2 to 40.9] | 36.7 [33.4 to 40.1]

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 to 1 Month After Dose 3
Description: An AE was any untoward medical occurrence in a participants, temporally associated with the use of study treatment, whether or not considered related to the study treatment. 95% CI was based on the Clopper and Pearson method. AEs reported in this outcome measure excluded local reactions and systemic events.
Time Frame: From Dose 1 to 1 Month after Dose 3
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. Here, 'Number of Participants Analyzed' = number of participants who received Dose 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 1001 | 987
Percentage of participants | 36.6 [33.6 to 39.6] | 39.4 [36.3 to 42.5]

10. Primary Outcome: Percentage of Participants With AEs From Dose 4 to 1 Month After Dose 4
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. 95% CI was based on the Clopper and Pearson method. AEs reported in this outcome measure excluded local reactions and systemic events.
Time Frame: From Dose 4 to 1 month after Dose 4
Population: Safety population included all the participants who received at least 1 dose of the IP with safety follow up after any dose. Here, 'Number of Participants Analyzed' = number of participants who received Dose 4 and had safety follow up after Dose 4.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 853 | 841
Percentage of participants | 15.1 [12.8 to 17.7] | 15.0 [12.6 to 17.6]

11. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 to 6 Months Following Dose 4
Description: A SAE was any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalisation or prolongation of existing hospitalisation; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect and other important medical events. 95% CI was based on the Clopper and Pearson method.
Time Frame: From Dose 1 to 6 months following Dose 4
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 1001 | 987
Percentage of participants | 4.5 [3.3 to 6.0] | 3.1 [2.1 to 4.4]

12. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Dose 1 to 6 Months Following Dose 4
Description: An NDCMC was defined as a significant disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects. 95% CI was based on the Clopper and Pearson method.
Time Frame: From Dose 1 to 6 months following Dose 4
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 1001 | 987
Percentage of participants | 5.0 [3.7 to 6.5] | 5.9 [4.5 to 7.5]

13. Primary Outcome: Percentage of Participants With Predefined Serotype-specific Immunoglobulin G (IgG) Concentrations 1 Month After Dose 3
Description: Pre-specified levels of serotypes were as follows: for serotype 1, 3, 4, 6A, 7F, 9V, 14, 18C, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, 33F: >=0.35 microgram per mL (mcg/mL), for serotype 5: >=0.23 mcg/mL, for serotype 6B: >=0.10 mcg/mL and for serotype 19A: >=0.12 mcg/mL. 95% CI was based on the Clopper and Pearson method.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population: eligible participants aged 42-98 days on Dose 1, received the first 3 doses randomized, had at least 1 valid immunogenicity result 27 to 56 days post Dose 3, and had no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population, "Number Analyzed" = number of participants with valid IgG concentrations for the specified serotype reported at 1 month after Dose 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 833 | 803
percentage of participants
  Serotype 1: number analyzed (Participants) | 833 | 802
  Serotype 1 | 79.8 [76.9 to 82.5] | 88.4 [86.0 to 90.5]
  Serotype 3: number analyzed (Participants) | 833 | 802
  Serotype 3 | 52.1 [48.6 to 55.5] | 67.6 [64.2 to 70.8]
  Serotype 4: number analyzed (Participants) | 833 | 802
  Serotype 4 | 79.7 [76.8 to 82.4] | 88.2 [85.7 to 90.3]
  Serotype 5: number analyzed (Participants) | 833 | 802
  Serotype 5 | 82.5 [79.7 to 85.0] | 86.8 [84.2 to 89.1]
  Serotype 6A: number analyzed (Participants) | 833 | 802
  Serotype 6A | 93.5 [91.6 to 95.1] | 95.9 [94.3 to 97.2]
  Serotype 6B: number analyzed (Participants) | 831 | 801
  Serotype 6B | 88.3 [85.9 to 90.4] | 92.4 [90.3 to 94.1]
  Serotype 7F: number analyzed (Participants) | 833 | 802
  Serotype 7F | 96.6 [95.2 to 97.8] | 97.6 [96.3 to 98.6]
  Serotype 9V: number analyzed (Participants) | 833 | 802
  Serotype 9V | 81.9 [79.1 to 84.4] | 89.8 [87.5 to 91.8]
  Serotype 14: number analyzed (Participants) | 832 | 802
  Serotype 14 | 93.4 [91.5 to 95.0] | 94.1 [92.3 to 95.7]
  Serotype 18C: number analyzed (Participants) | 833 | 802
  Serotype 18C | 92.6 [90.6 to 94.2] | 93.1 [91.2 to 94.8]
  Serotype 19A: number analyzed (Participants) | 833 | 802
  Serotype 19A | 97.1 [95.7 to 98.1] | 98.1 [96.9 to 98.9]
  Serotype 19F: number analyzed (Participants) | 833 | 802
  Serotype 19F | 96.9 [95.5 to 98.0] | 96.6 [95.1 to 97.8]
  Serotype 23F: number analyzed (Participants) | 833 | 802
  Serotype 23F | 77.9 [74.9 to 80.7] | 85.5 [82.9 to 87.9]
  Serotype 8 | 96.8 [95.3 to 97.9] | 85.5 [82.9 to 87.9]
  Serotype 10A | 82.2 [79.5 to 84.8] | 85.5 [82.9 to 87.9]
  Serotype 11A | 92.7 [90.7 to 94.4] | 85.5 [82.9 to 87.9]
  Serotype 12F | 67.5 [64.2 to 70.6] | 85.5 [82.9 to 87.9]
  Serotype 15B | 98.2 [97.0 to 99.0] | 85.5 [82.9 to 87.9]
  Serotype 22F | 98.3 [97.2 to 99.1] | 85.5 [82.9 to 87.9]
  Serotype 33F: number analyzed (Participants) | 833 | 802
  Serotype 33F | 86.7 [84.2 to 88.9] | 85.5 [82.9 to 87.9]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Serotype 1: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — Comparison was conducted for the 13 matched serotypes for 20vPnC to the corresponding serotype in 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the percentage differences (20vPnC - 13vPnC) was greater than -10%; percentage difference = -8.6, 95% CI 2-sided [-12.1 to -5.1]
Statistical Analysis 2: Comparison: 20vPnC vs 13vPnC; Serotype 3: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -15.5, 95% CI 2-sided [-20.1 to -10.8]
Statistical Analysis 3: Comparison: 20vPnC vs 13vPnC; Serotype 4: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -8.4, 95% CI 2-sided [-12.0 to -4.9]
Statistical Analysis 4: Comparison: 20vPnC vs 13vPnC; Serotype 5: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -4.3, 95% CI 2-sided [-7.8 to -0.8]
Statistical Analysis 5: Comparison: 20vPnC vs 13vPnC; Serotype 6A: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -2.4, 95% CI 2-sided [-4.6 to -0.2]
Statistical Analysis 6: Comparison: 20vPnC vs 13vPnC; Serotype 6B: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -4.1, 95% CI 2-sided [-7.0 to -1.2]
Statistical Analysis 7: Comparison: 20vPnC vs 13vPnC; Serotype 7F: 2-sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -1.0, 95% CI 2-sided [-2.7 to 0.7]
Statistical Analysis 8: Comparison: 20vPnC vs 13vPnC; Serotype 9V: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -7.9, 95% CI 2-sided [-11.3 to -4.6]
Statistical Analysis 9: Comparison: 20vPnC vs 13vPnC; Serotype 14: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -0.8, 95% CI 2-sided [-3.1 to 1.6]
Statistical Analysis 10: Comparison: 20vPnC vs 13vPnC; Serotype 18C: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -0.6, 95% CI 2-sided [-3.1 to 1.9]
Statistical Analysis 11: Comparison: 20vPnC vs 13vPnC; Serotype 19A: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -1.0, 95% CI 2-sided [-2.6 to 0.5]
Statistical Analysis 12: Comparison: 20vPnC vs 13vPnC; Serotype 19F: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = 0.2, 95% CI 2-sided [-1.5 to 2.0]
Statistical Analysis 13: Comparison: 20vPnC vs 13vPnC; Serotype 23F: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; percentage difference = -7.6, 95% CI 2-sided [-11.4 to -3.9]
Statistical Analysis 14: Comparison: 20vPnC vs 13vPnC; Serotype 8: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results were from serotype 23F (13vPnC serotype with the lowest percentage, not including serotype 3) in the 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the percentage differences (20vPnC - lowest 13vPnC) was greater than -10%; percentage difference = 11.2, 95% CI 2-sided [8.6 to 14.0]
Statistical Analysis 15: Comparison: 20vPnC vs 13vPnC; Serotype 10A: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; percentage difference = -3.3, 95% CI 2-sided [-6.9 to 0.3]
Statistical Analysis 16: Comparison: 20vPnC vs 13vPnC; Serotype 11A: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; percentage difference = 7.1, 95% CI [4.2 to 10.2]
Statistical Analysis 17: Comparison: 20vPnC vs 13vPnC; Serotype 12F: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; percentage difference = -18.1, 95% CI 2-sided [-22.1 to -14.0]
Statistical Analysis 18: Comparison: 20vPnC vs 13vPnC; Serotype 15B: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; percentage difference = 12.7, 95% CI 2-sided [10.2 to 15.4]
Statistical Analysis 19: Comparison: 20vPnC vs 13vPnC; Serotype 22F: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; percentage difference = 12.8, 95% CI 2-sided [10.3 to 15.5]
Statistical Analysis 20: Comparison: 20vPnC vs 13vPnC; Serotype 33F: 2-Sided CI were calculated based on the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 14]; percentage difference = 1.1, 95% CI 2-sided [-2.2 to 4.5]

14. Primary Outcome: Serotype-specific IgG Geometric Mean Concentration (GMCs) and Geometric Mean Ratios (GMRs) at 1 Month After Dose 4
Description: Concentrations of anticapsular IgG for the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, and 33F) were determined in all participants at 1 month after Dose 4 using the Luminex assay. Results were expressed as IgG concentrations. GMCs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution. Assay result below LLOQ was set to 0.5*LLOQ. Geometric mean ratios (GMRs) were reported in statistical analysis section and were calculated by exponentiating mean difference of logarithm of concentration and corresponding 2-sided 95% CIs (based on Student's t distribution).
Time Frame: From Dose 1 to 6 months following Dose 4
Population: Dose 4 evaluable immunogenicity population: aged 42-98 days on Dose 1, received the first 4 doses randomized, had at least 1 valid immunogenicity result 27 to 56 days after Dose 4, had no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 4 evaluable immunogenicity population, "Number Analyzed" = number of participants with valid IgG concentrations for the specified serotype reported at 1 month after Dose 4.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (μg/mL)
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 755 | 745
microgram per milliliter (μg/mL)
  Serotype 1: number analyzed (Participants) | 755 | 744
  Serotype 1 | 1.47 [1.37 to 1.57] | 2.12 [1.97 to 2.27]
  Serotype 3 | 0.56 [0.53 to 0.60] | 0.85 [0.80 to 0.90]
  Serotype 4: number analyzed (Participants) | 754 | 745
  Serotype 4 | 3.77 [3.52 to 4.04] | 4.84 [4.50 to 5.22]
  Serotype 5 | 1.87 [1.74 to 2.00] | 2.51 [2.33 to 2.70]
  Serotype 6A | 9.01 [8.45 to 9.61] | 11.69 [10.91 to 12.53]
  Serotype 6B: number analyzed (Participants) | 753 | 744
  Serotype 6B | 4.01 [3.70 to 4.35] | 5.74 [5.27 to 6.24]
  Serotype 7F | 3.91 [3.70 to 4.35] | 5.18 [4.88 to 5.49]
  Serotype 9V: number analyzed (Participants) | 755 | 744
  Serotype 9V | 3.44 [3.23 to 3.67] | 4.30 [4.02 to 4.59]
  Serotype 14 | 5.68 [5.27 to 6.12] | 6.34 [5.88 to 6.83]
  Serotype 18C | 3.46 [3.24 to 3.70] | 4.69 [4.34 to 5.05]
  Serotype 19A: number analyzed (Participants) | 754 | 745
  Serotype 19A | 3.53 [3.30 to 3.77] | 4.13 [3.84 to 4.45]
  Serotype 19F | 5.01 [4.68 to 5.36] | 5.79 [5.36 to 6.25]
  Serotype 23F | 3.95 [3.63 to 4.31] | 6.18 [5.66 to 6.75]
  Serotype 8: number analyzed (Participants) | 755 | 720
  Serotype 8 | 3.97 [3.73 to 4.22] | 0.03 [0.03 to 0.04]
  Serotype 10A | 6.22 [5.75 to 6.72] | 0.01 [0.01 to 0.01]
  Serotype 11A | 3.53 [3.31 to 3.78] | 0.02 [0.02 to 0.02]
  Serotype 12F | 1.85 [1.73 to 1.99] | 0.01 [0.01 to 0.01]
  Serotype 15B | 12.59 [11.78 to 13.45] | 0.02 [0.02 to 0.03]
  Serotype 22F | 10.60 [9.92 to 11.33] | 0.00 [0.00 to 0.01]
  Serotype 33F | 9.31 [8.71 to 9.96] | 0.01 [0.01 to 0.01]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Serotype 1: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC was to the corresponding serotype in 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the IgG GMR of 20vPnC to 13vPnC for the serotype is greater than 0.5 (2-fold NI margin); Geometric Mean Ratio = 0.69, 95% CI 2-sided [0.63 to 0.76]
Statistical Analysis 2: Comparison: 20vPnC vs 13vPnC; Serotype 3: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.66, 95% CI 2-sided [0.61 to 0.73]
Statistical Analysis 3: Comparison: 20vPnC vs 13vPnC; Serotype 4: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.78, 95% CI [0.70 to 0.86]
Statistical Analysis 4: Comparison: 20vPnC vs 13vPnC; Serotype 5: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.74, 95% CI 2-sided [0.67 to 0.82]
Statistical Analysis 5: Comparison: 20vPnC vs 13vPnC; Serotype 6A: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.70 to 0.85]
Statistical Analysis 6: Comparison: 20vPnC vs 13vPnC; Serotype 6B: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.70, 95% CI 2-sided [0.62 to 0.79]
Statistical Analysis 7: Comparison: 20vPnC vs 13vPnC; Serotype 7F: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.76, 95% CI 2-sided [0.70 to 0.82]
Statistical Analysis 8: Comparison: 20vPnC vs 13vPnC; Serotype 9V: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.80, 95% CI [0.73 to 0.88]
Statistical Analysis 9: Comparison: 20vPnC vs 13vPnC; Serotype 14: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.90, 95% CI 2-sided [0.81 to 1.00]
Statistical Analysis 10: Comparison: 20vPnC vs 13vPnC; Serotype 18C: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.74, 95% CI [0.67 to 0.82]
Statistical Analysis 11: Comparison: 20vPnC vs 13vPnC; Serotype 19A: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.85, 95% CI 2-sided [0.77 to 0.94]
Statistical Analysis 12: Comparison: 20vPnC vs 13vPnC; Serotype 19F: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.86, 95% CI 2-sided [0.78 to 0.96]
Statistical Analysis 13: Comparison: 20vPnC vs 13vPnC; Serotype 23F: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC-13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 1]; Geometric Mean Ratio = 0.64, 95% CI 2-sided [0.57 to 0.72]
Statistical Analysis 14: Comparison: 20vPnC vs 13vPnC; Serotype 8: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — For the additional 7 serotypes, the compared results were from serotype 1 (13vPnC serotype with the lowest GMC, not including serotype 3) in the 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC/lowest 13vPnC) was greater than 0.5 (2-fold criterion); Geometric Mean Ratio = 1.87, 95% CI 2-sided [1.71 to 2.06]
Statistical Analysis 15: Comparison: 20vPnC vs 13vPnC; Serotype 10A: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; Geometric Mean Ratio = 2.94, 95% CI [2.64 to 3.26]
Statistical Analysis 16: Comparison: 20vPnC vs 13vPnC; Serotype 11A: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; Geometric Mean Ratio = 1.67, 95% CI 2-sided [1.51 to 1.84]
Statistical Analysis 17: Comparison: 20vPnC vs 13vPnC; Serotype 12F: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; Geometric Mean Ratio = 0.88, 95% CI [0.79 to 0.97]
Statistical Analysis 18: Comparison: 20vPnC vs 13vPnC; Serotype 15B: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; Geometric Mean Ratio = 5.95, 95% CI [5.39 to 6.55]
Statistical Analysis 19: Comparison: 20vPnC vs 13vPnC; Serotype 22F: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; Geometric Mean Ratio = 5.01, 95% CI [4.54 to 5.52]
Statistical Analysis 20: Comparison: 20vPnC vs 13vPnC; Serotype 33F: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - lowest 13vPnC) of the logarithms of the IgG concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 14, analysis 14]; Geometric Mean Ratio = 4.40, 95% CI 2-sided [3.99 to 4.85]

15. Primary Outcome: Percentage of Participants With Prespecified Antibody Levels to Specific Concomitant Vaccine Antigens 1 Month After Dose 3
Description: Concentration of antibody to diphtheria toxoid (predefined level ≥0.1 IU/mL), tetanus toxoid (predefined level ≥0.1 IU/mL), IgG antibodies to pertussis antigens (pertussis toxin, filamentous hemagglutinin and pertactin, each with the predefined level as the 5th percentile observed in the 13vPnC group), hepatitis B antibody (in milli-international units per mL [mIU/mL]) (predefined level ≥10 mIU/mL), neutralizing antibody (NA) titers to poliovirus types 1, 2, and 3 (predefined level NA titer ≥1:8), Haemophilus influenzae type b (Hib) (≥0.15 μg/mL) were determined on subsets of sera collected at the immunogenicity time point 1 month after Dose 3. The antibody levels were measured by a validated multiplex Luminex immunoassay. The concomitant immune responses were measured on random subsets.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable population: eligible participants aged 42-98 days on Dose 1, received the first 3 doses randomized, had at least 1 valid immunogenicity result 27 to 56 days post Dose 3, had no major protocol deviations. "Number of Participants Analyzed"=participants in Dose 3 evaluable immunogenicity population, "Number Analyzed" = number of participants with valid assay results for the specified antigen at 1 month after Dose 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 833 | 803
percentage of participants
  Diphtheria: number analyzed (Participants) | 370 | 363
  Diphtheria | 93.5 [90.5 to 95.8] | 97.8 [95.7 to 99.0]
  Tetanus: number analyzed (Participants) | 370 | 363
  Tetanus | 99.7 [98.5 to 100.0] | 99.4 [98.0 to 99.9]
  Pertussis (PT): number analyzed (Participants) | 370 | 363
  Pertussis (PT) | 94.9 [92.1 to 96.9] | 95.0 [92.3 to 97.0]
  Pertussis (FHA): number analyzed (Participants) | 370 | 363
  Pertussis (FHA) | 95.7 [93.1 to 97.5] | 95.0 [92.3 to 97.0]
  Pertussis (PRN): number analyzed (Participants) | 370 | 363
  Pertussis (PRN) | 93.8 [90.8 to 96.0] | 95.0 [92.3 to 97.0]
  hepatitis B surface antigen (HBsAg): number analyzed (Participants) | 118 | 127
  hepatitis B surface antigen (HBsAg) | 100.0 [96.9 to 100.0] | 100.0 [97.1 to 100.0]
  Poliovirus (Type 1): number analyzed (Participants) | 111 | 117
  Poliovirus (Type 1) | 100.0 [96.7 to 100.0] | 100.0 [96.9 to 100.0]
  Poliovirus (Type 2): number analyzed (Participants) | 115 | 120
  Poliovirus (Type 2) | 100.0 [96.8 to 100.0] | 99.2 [95.4 to 100.0]
  Poliovirus (Type 3): number analyzed (Participants) | 115 | 120
  Poliovirus (Type 3) | 100.0 [96.8 to 100.0] | 100.0 [97.0 to 100.0]
  Hib ≥0.15 μg/mL: number analyzed (Participants) | 124 | 125
  Hib ≥0.15 μg/mL | 100.0 [97.1 to 100.0] | 100.0 [97.1 to 100.0]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Diphtheria: 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CI for the percentage differences (20vPnC - 13vPnC) was greater than -10%; Percentage Difference = -4.3, 95% CI 2-sided [-7.5 to -1.4]
Statistical Analysis 2: Comparison: 20vPnC vs 13vPnC; Tetanus: 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.3, 95% CI 2-sided [-1.0 to 1.7]
Statistical Analysis 3: Comparison: 20vPnC vs 13vPnC; Pertussis (PT): 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = -0.2, 95% CI [-3.5 to 3.1]
Statistical Analysis 4: Comparison: 20vPnC vs 13vPnC; Pertussis (FHA): 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.6, 95% CI [-2.5 to 3.9]
Statistical Analysis 5: Comparison: 20vPnC vs 13vPnC; Pertussis (PRN): 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage.2-Sided CIs are calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = -1.3, 95% CI [-4.7 to 2.2]
Statistical Analysis 6: Comparison: 20vPnC vs 13vPnC; HBsAg: 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.0, 95% CI [-3.2 to 2.9]
Statistical Analysis 7: Comparison: 20vPnC vs 13vPnC; Poliovirus (Type 1): 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.0, 95% CI [-3.4 to 3.2]
Statistical Analysis 8: Comparison: 20vPnC vs 13vPnC; Poliovirus (Type 2): 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.8, 95% CI [-2.4 to 4.6]
Statistical Analysis 9: Comparison: 20vPnC vs 13vPnC; Poliovirus (Type 3): 2-Sided CI was calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.0, 95% CI [-3.2 to 3.1]
Statistical Analysis 10: Comparison: 20vPnC vs 13vPnC; Hib (≥0.15 μg/mL): 2-Sided CI were calculated using the Miettinen and Nurminen method for the difference in proportions, expressed as a percentage; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; Percentage Difference = 0.0, 95% CI 2-sided [-3.0 to 3.0]

16. Secondary Outcome: Serotype-specific IgG GMCs and GMRs at 1 Month After Dose 3
Description: Pneumococcal IgG antibody against each of the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F) was measured using direct binding Luminex assay. Results were expressed as IgG concentrations. GMCs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution. Assay result below LLOQ were set to 0.5*LLOQ.GMRs were reported in statistical analysis section and were calculated by exponentiating mean difference of logarithm of concentration and corresponding 2-sided 95% CI (based on Student's t distribution). Assay result below LLOQ were set to 0.5*LLOQ.GMRs were reported in statistical analysis section and were calculated by exponentiating mean difference of logarithm of concentration and corresponding 2-sided 95% CI (based on Student's t distribution).
Time Frame: 1 month after Dose 3
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 833 | 803
μg/mL
  Serotype 1: number analyzed (Participants) | 833 | 802
  Serotype 1 | 0.74 [0.70 to 0.79] | 1.14 [1.06 to 1.22]
  Serotype 3: number analyzed (Participants) | 833 | 802
  Serotype 3 | 0.36 [0.33 to 0.38] | 0.51 [0.48 to 0.55]
  Serotype 4: number analyzed (Participants) | 833 | 802
  Serotype 4 | 0.75 [0.70 to 0.81] | 1.08 [1.00 to 1.17]
  Serotype 5: number analyzed (Participants) | 833 | 802
  Serotype 5 | 0.66 [0.61 to 0.71] | 0.96 [0.88 to 1.04]
  Serotype 6A: number analyzed (Participants) | 833 | 802
  Serotype 6A | 1.95 [1.81 to 2.10] | 2.69 [2.48 to 2.92]
  Serotype 6B: number analyzed (Participants) | 831 | 801
  Serotype 6B | 0.61 [0.55 to 0.68] | 1.02 [0.91 to 1.14]
  Serotype 7F: number analyzed (Participants) | 833 | 802
  Serotype 7F | 1.71 [1.62 to 1.81] | 2.29 [2.16 to 2.43]
  Serotype 9V: number analyzed (Participants) | 833 | 802
  Serotype 9V | 0.87 [0.81 to 0.93] | 1.21 [1.12 to 1.30]
  Serotype 14: number analyzed (Participants) | 832 | 802
  Serotype 14 | 2.16 [2.01 to 2.33] | 2.72 [2.51 to 2.95]
  Serotype 18C: number analyzed (Participants) | 833 | 802
  Serotype 18C | 1.31 [1.23 to 1.39] | 1.71 [1.59 to 1.84]
  Serotype 19A: number analyzed (Participants) | 833 | 802
  Serotype 19A | 0.72 [0.67 to 0.76] | 0.91 [0.85 to 0.97]
  Serotype 19F: number analyzed (Participants) | 833 | 802
  Serotype 19F | 1.59 [1.50 to 1.67] | 2.00 [1.88 to 2.12]
  Serotype 23F: number analyzed (Participants) | 833 | 802
  Serotype 23F | 0.82 [0.75 to 0.90] | 1.25 [1.14 to 1.37]
  Serotype 8: number analyzed (Participants) | 833 | 794
  Serotype 8 | 1.80 [1.70 to 1.91] | 0.02 [0.02 to 0.02]
  Serotype 10A | 1.21 [1.09 to 1.33] | 0.01 [0.01 to 0.01]
  Serotype 11A | 1.39 [1.30 to 1.48] | 0.02 [0.01 to 0.02]
  Serotype 12F | 0.55 [0.50 to 0.60] | 0.01 [0.01 to 0.01]
  Serotype 15B | 4.40 [4.11 to 4.71] | 0.03 [0.02 to 0.03]
  Serotype 22F | 3.71 [3.45 to 3.99] | 0.01 [0.00 to 0.01]
  Serotype 33F: number analyzed (Participants) | 833 | 802
  Serotype 33F | 1.49 [1.36 to 1.64] | 0.02 [0.01 to 0.02]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 1]; Test type: Non-Inferiority — Comparison for the 13 matched serotypes for 20vPnC is to the corresponding serotype in 13vPnC group. Noninferiority was declared for if the lower bound of the 2-sided 95% CI for the IgG GMR of 20vPnC to 13vPnC for the serotype is greater than 0.5 (2-fold NI margin); Geometric Mean Ratios = 0.65, 95% CI 2-sided [0.59 to 0.72]
Statistical Analysis 2: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.70, 95% CI 2-sided [0.64 to 0.76]
Statistical Analysis 3: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 3]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.70, 95% CI [0.63 to 0.78]
Statistical Analysis 4: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 4]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.69, 95% CI [0.61 to 0.77]
Statistical Analysis 5: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 5]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.72, 95% CI [0.65 to 0.81]
Statistical Analysis 6: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 6]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.51 to 0.70]
Statistical Analysis 7: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 7]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.75, 95% CI [0.69 to 0.81]
Statistical Analysis 8: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 8]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.72, 95% CI 2-sided [0.65 to 0.80]
Statistical Analysis 9: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 9]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.79, 95% CI [0.71 to 0.89]
Statistical Analysis 10: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 10]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.77, 95% CI [0.70 to 0.84]
Statistical Analysis 11: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 11]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.79, 95% CI 2-sided [0.72 to 0.86]
Statistical Analysis 12: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 12]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.79, 95% CI [0.73 to 0.86]
Statistical Analysis 13: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 13]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 1]; Geometric Mean Ratio = 0.66, 95% CI 2-sided [0.58 to 0.75]
Statistical Analysis 14: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 14]; Test type: Non-Inferiority — For the additional 7 serotypes, the compared results are from serotype 19A (13vPnC serotype with the lowest GMC, not including serotype 3) in the 13vPnC group. Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (20vPnC/lowest 13vPnC) was greater than 0.5 (2-fold criterion); Geometric Mean Ratio = 1.98, 95% CI [1.81 to 2.16]
Statistical Analysis 15: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 15]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 14]; Geometric Mean Ratio = 1.32, 95% CI [1.18 to 1.49]
Statistical Analysis 16: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 16]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 14]; Geometric Mean Ratio = 1.52, 95% CI [1.39 to 1.67]
Statistical Analysis 17: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 17]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 14]; Geometric Mean Ratio = 0.60, 95% CI [0.54 to 0.67]
Statistical Analysis 18: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 18]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 14]; Geometric Mean Ratio = 4.82, 95% CI 2-sided [4.39 to 5.30]
Statistical Analysis 19: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 19]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 14]; Geometric Mean Ratio = 4.06, 95% CI [3.68 to 4.48]
Statistical Analysis 20: Comparison: 20vPnC vs 13vPnC; [analysis description as in outcome 14, analysis 20]; Test type: Non-Inferiority — [test comment as in outcome 16, analysis 14]; Geometric Mean Ratio = 1.64, 95% CI [1.46 to 1.83]

17. Secondary Outcome: Percentage of Participants With Predefined IgG Concentrations 1 Month After Dose 4
Description: as for outcome 13
Time Frame: 1 month after Dose 4
Population: Dose 4 evaluable immunogenicity population: eligible participants aged 42-98 days on Dose 1, received all 4 doses as randomized, had at least 1 valid immunogenicity result within 27 to 56 days after Dose 4, and had no other major protocol deviations. "Number of Participants Analyzed"=participants in Dose 4 evaluable immunogenicity population, "Number Analyzed" = number of participants with valid IgG concentrations for the specified serotype reported at 1 month after Dose 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 755 | 745
percentage of participants
  Serotype 1: number analyzed (Participants) | 755 | 744
  Serotype 1 | 94.3 [92.4 to 95.8] | 97.2 [95.7 to 98.2]
  Serotype 3 | 73.6 [70.3 to 76.8] | 85.8 [83.1 to 88.2]
  Serotype 4: number analyzed (Participants) | 754 | 745
  Serotype 4 | 98.9 [97.9 to 99.5] | 99.1 [98.1 to 99.6]
  Serotype 5 | 97.9 [96.6 to 98.8] | 97.7 [96.4 to 98.7]
  Serotype 6A | 99.5 [98.6 to 99.9] | 99.7 [99.0 to 100.0]
  Serotype 6B: number analyzed (Participants) | 753 | 744
  Serotype 6B | 99.1 [98.1 to 99.6] | 99.5 [98.6 to 99.9]
  Serotype 7F | 99.5 [98.6 to 99.9] | 99.9 [99.3 to 100.0]
  Serotype 9V: number analyzed (Participants) | 755 | 744
  Serotype 9V | 98.5 [97.4 to 99.3] | 98.9 [97.9 to 99.5]
  Serotype 14 | 98.9 [97.9 to 99.5] | 99.5 [98.6 to 99.9]
  Serotype 18C | 98.9 [97.9 to 99.5] | 99.5 [98.6 to 99.9]
  Serotype 19A: number analyzed (Participants) | 754 | 745
  Serotype 19A | 99.9 [99.3 to 100.0] | 99.7 [99.0 to 100.0]
  Serotype 19F | 98.8 [97.7 to 99.5] | 98.9 [97.9 to 99.5]
  Serotype 23F | 97.2 [95.8 to 98.3] | 98.1 [96.9 to 99.0]
  Serotype 8: number analyzed (Participants) | 755 | 744
  Serotype 8 | 99.5 [98.6 to 99.9] | 4.7 [3.3 to 6.5]
  Serotype 10A: number analyzed (Participants) | 755 | 744
  Serotype 10A | 97.7 [96.4 to 98.7] | 2.0 [1.1 to 3.3]
  Serotype 11A: number analyzed (Participants) | 755 | 744
  Serotype 11A | 98.8 [97.7 to 99.5] | 4.2 [2.8 to 5.9]
  Serotype 12F: number analyzed (Participants) | 755 | 744
  Serotype 12F | 95.2 [93.5 to 96.6] | 0.3 [0.0 to 1.0]
  Serotype 15B: number analyzed (Participants) | 755 | 744
  Serotype 15B | 99.7 [99.0 to 100.0] | 4.6 [3.2 to 6.3]
  Serotype 22F: number analyzed (Participants) | 755 | 744
  Serotype 22F | 99.6 [98.8 to 99.9] | 1.5 [0.7 to 2.6]
  Serotype 33F: number analyzed (Participants) | 755 | 744
  Serotype 33F | 99.5 [98.6 to 99.9] | 1.7 [0.9 to 3.0]

18. Secondary Outcome: Serotype-Specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at 1 Month After Dose 3
Description: OPA titers for the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, and 33F) were determined in randomized subsets of participants at 1 month after Dose 3. Results were expressed as OPA titers. GMTs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution. OPA titers were determined in randomized subsets of participants at 1 month after Dose 3.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable immunogenicity population: aged 42-98 days on Dose 1, received the first 3 doses randomized, had at least 1 valid immunogenicity result 27 to 56 days after Dose 3, had no protocol deviations. "Number of Participants Analyzed" = Dose 3 evaluable immunogenicity populations. "Number Analyzed" = number of participants with valid OPA titers for the specified serotype reported at 1 month after Dose 3.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 833 | 803
Titers
  Serotype 1: number analyzed (Participants) | 103 | 98
  Serotype 1 | 26 [21 to 33] | 34 [27 to 42]
  Serotype 3: number analyzed (Participants) | 105 | 97
  Serotype 3 | 51 [43 to 61] | 63 [53 to 76]
  Serotype 4: number analyzed (Participants) | 97 | 90
  Serotype 4 | 339 [252 to 455] | 280 [207 to 378]
  Serotype 5: number analyzed (Participants) | 103 | 98
  Serotype 5 | 32 [27 to 39] | 39 [32 to 47]
  Serotype 6A: number analyzed (Participants) | 104 | 96
  Serotype 6A | 910 [763 to 1084] | 936 [757 to 1156]
  Serotype 6B: number analyzed (Participants) | 99 | 91
  Serotype 6B | 318 [242 to 419] | 516 [409 to 651]
  Serotype 7F: number analyzed (Participants) | 91 | 87
  Serotype 7F | 1222 [1020 to 1465] | 1149 [926 to 1424]
  Serotype 9V: number analyzed (Participants) | 94 | 87
  Serotype 9V | 661 [482 to 906] | 594 [421 to 838]
  Serotype 14: number analyzed (Participants) | 103 | 97
  Serotype 14 | 415 [323 to 535] | 420 [330 to 535]
  Serotype 18C: number analyzed (Participants) | 95 | 87
  Serotype 18C | 1153 [910 to 1460] | 996 [754 to 1317]
  Serotype 19A: number analyzed (Participants) | 93 | 84
  Serotype 19A | 108 [78 to 149] | 109 [79 to 151]
  Serotype 19F: number analyzed (Participants) | 102 | 97
  Serotype 19F | 84 [67 to 105] | 116 [90 to 149]
  Serotype 23F: number analyzed (Participants) | 96 | 86
  Serotype 23F | 255 [186 to 350] | 295 [215 to 406]
  Serotype 8: number analyzed (Participants) | 100 | 112
  Serotype 8 | 665 [503 to 880] | 18 [17 to 20]
  Serotype 10A: number analyzed (Participants) | 101 | 109
  Serotype 10A | 2558 [1869 to 3501] | 37 [33 to 42]
  Serotype 11A: number analyzed (Participants) | 100 | 108
  Serotype 11A | 289 [212 to 395] | 50 [46 to 55]
  Serotype 12F: number analyzed (Participants) | 92 | 110
  Serotype 12F | 7677 [5952 to 9901] | 28 [24 to 33]
  Serotype 15B: number analyzed (Participants) | 97 | 110
  Serotype 15B | 1560 [1090 to 2233] | 18 [16 to 22]
  Serotype 22F: number analyzed (Participants) | 97 | 113
  Serotype 22F | 6797 [5170 to 8936] | 9 [9 to 9]
  Serotype 33F: number analyzed (Participants) | 85 | 111
  Serotype 33F | 7388 [4803 to 11365] | 198 [177 to 220]

19. Secondary Outcome: Serotype-specific OPA GMTs at 1 Month After Dose 4
Description: OPA titers for the 20 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F, and 33F) were determined in randomized subsets of participants at 1 month after Dose 4. Results were expressed as OPA titers. GMTs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution. OPA titers were determined in randomized subsets of participants at 1 month after Dose 4.
Time Frame: 1 month after Dose 4
Population: Dose 4 evaluable immunogenicity population: aged 42-98 days on Dose 1, received the first 4 doses randomized, had at least 1 valid immunogenicity result 27 to 56 days after Dose 4, had no major protocol deviations. "Number of Participants Analyzed" = Dose 4 evaluable immunogenicity populations. "Number Analyzed" = number of participants with valid OPA titers for the specified serotype reported at 1 month after Dose 4.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 755 | 745
Titers
  Serotype 1: number analyzed (Participants) | 94 | 91
  Serotype 1 | 36 [27 to 48] | 66 [50 to 87]
  Serotype 3: number analyzed (Participants) | 92 | 88
  Serotype 3 | 62 [49 to 78] | 102 [86 to 120]
  Serotype 4: number analyzed (Participants) | 85 | 82
  Serotype 4 | 621 [435 to 887] | 961 [714 to 1294]
  Serotype 5: number analyzed (Participants) | 94 | 91
  Serotype 5 | 55 [45 to 67] | 69 [54 to 87]
  Serotype 6A: number analyzed (Participants) | 93 | 91
  Serotype 6A | 1384 [1092 to 1753] | 1767 [1329 to 2348]
  Serotype 6B: number analyzed (Participants) | 92 | 88
  Serotype 6B | 666 [489 to 906] | 1211 [861 to 1703]
  Serotype 7F: number analyzed (Participants) | 84 | 81
  Serotype 7F | 2022 [1673 to 2444] | 2099 [1741 to 2531]
  Serotype 9V: number analyzed (Participants) | 85 | 79
  Serotype 9V | 2609 [1913 to 3558] | 3210 [2500 to 4123]
  Serotype 14: number analyzed (Participants) | 92 | 91
  Serotype 14 | 667 [523 to 850] | 593 [462 to 761]
  Serotype 18C: number analyzed (Participants) | 84 | 83
  Serotype 18C | 1973 [1472 to 2643] | 2425 [1914 to 3072]
  Serotype 19A: number analyzed (Participants) | 85 | 78
  Serotype 19A | 844 [622 to 1145] | 1357 [1007 to 1829]
  Serotype 19F: number analyzed (Participants) | 93 | 91
  Serotype 19F | 246 [179 to 337] | 373 [272 to 513]
  Serotype 23F: number analyzed (Participants) | 84 | 77
  Serotype 23F | 827 [554 to 1235] | 1532 [1118 to 2100]
  Serotype 8: number analyzed (Participants) | 89 | 97
  Serotype 8 | 1228 [901 to 1673] | 26 [21 to 31]
  Serotype 10A: number analyzed (Participants) | 99 | 102
  Serotype 10A | 3674 [2746 to 4916] | 57 [44 to 74]
  Serotype 11A: number analyzed (Participants) | 90 | 89
  Serotype 11A | 2728 [1975 to 3768] | 69 [53 to 89]
  Serotype 12F: number analyzed (Participants) | 86 | 103
  Serotype 12F | 9320 [7037 to 12343] | 31 [26 to 37]
  Serotype 15B: number analyzed (Participants) | 92 | 100
  Serotype 15B | 3035 [2138 to 4308] | 23 [17 to 30]
  Serotype 22F: number analyzed (Participants) | 86 | 101
  Serotype 22F | 11077 [7956 to 15422] | 15 [11 to 20]
  Serotype 33F: number analyzed (Participants) | 80 | 97
  Serotype 33F | 19216 [13193 to 27990] | 363 [292 to 451]

20. Secondary Outcome: Serotype-specific IgG Geometric Mean Fold Rise (GMFRs) From 1 Month After Dose 3 to Before Dose 4
Description: GMFR of pneumococcal 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F and 33F. The GMFR from 1 month after Dose 3 to before Dose 4 were reported from Dose 3 evaluable immunogenicity participant.
Time Frame: 1 month after Dose 3 to before Dose 4
Population: Dose 3 evaluable immunogenicity population: eligible participants aged 42-98 days on Dose 1, received the first 3 doses as randomized, had at least 1 valid immunogenicity result 27 to 56 days after Dose 3, and had no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 3 evaluable immunogenicity population; "Number Analyzed"= number of participants with valid IgG concentrations at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 758 | 733
Fold rise
  Serotype 1 | 0.3 [0.3 to 0.3] | 0.3 [0.2 to 0.3]
  Serotype 3 | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]
  Serotype 4 | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.3]
  Serotype 5 | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.3]
  Serotype 6A: number analyzed (Participants) | 758 | 732
  Serotype 6A | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.3]
  Serotype 6B: number analyzed (Participants) | 754 | 730
  Serotype 6B | 0.4 [0.4 to 0.4] | 0.3 [0.3 to 0.3]
  Serotype 7F | 0.4 [0.4 to 0.6] | 0.4 [0.3 to 0.4]
  Serotype 9V | 0.3 [0.3 to 0.4] | 0.3 [0.3 to 0.3]
  Serotype 14: number analyzed (Participants) | 757 | 733
  Serotype 14 | 0.5 [0.4 to 0.5] | 0.5 [0.4 to 0.5]
  Serotype 18C | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]
  Serotype 19A: number analyzed (Participants) | 757 | 733
  Serotype 19A | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2]
  Serotype 19F | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.2]
  Serotype 23F | 0.3 [0.3 to 0.3] | 0.3 [0.2 to 0.3]
  Serotype 8: number analyzed (Participants) | 758 | 706
  Serotype 8 | 0.2 [0.2 to 0.3] | 1.4 [1.3 to 1.5]
  Serotype 10A: number analyzed (Participants) | 758 | 732
  Serotype 10A | 0.7 [0.6 to 0.7] | 0.9 [0.9 to 1.0]
  Serotype 11A: number analyzed (Participants) | 758 | 732
  Serotype 11A | 0.3 [0.2 to 0.3] | 1.1 [1.0 to 1.2]
  Serotype 12F: number analyzed (Participants) | 758 | 732
  Serotype 12F | 0.3 [0.3 to 0.4] | 1.0 [1.0 to 1.1]
  Serotype 15B: number analyzed (Participants) | 758 | 732
  Serotype 15B | 0.4 [0.3 to 0.4] | 0.8 [0.7 to 0.8]
  Serotype 22F: number analyzed (Participants) | 758 | 732
  Serotype 22F | 0.3 [0.3 to 0.4] | 0.8 [0.7 to 0.9]
  Serotype 33F: number analyzed (Participants) | 758 | 731
  Serotype 33F | 0.7 [0.7 to 0.8] | 0.8 [0.7 to 0.8]

21. Secondary Outcome: Serotype-specific IgG GMFRs From 1 Month Before to 1 Month After Dose 4
Description: GMFR of pneumococcal 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F and 33F. The GMFR from 1 month before Dose 4 to 1 month after Dose 4 were reported from Dose 4 evaluable immunogenicity participants.
Time Frame: From 1 month before to 1 month after Dose 4
Population: Dose 4 evaluable immunogenicity population: eligible participants aged 42-98 days on Dose 1, received all 4 doses as randomized, had at least 1 valid immunogenicity result 27 to 56 days after Dose 4, and had no major protocol deviations. "Number of Participants Analyzed"= participants in Dose 4 evaluable immunogenicity population; "Number Analyzed"= number of participants with valid IgG concentrations at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 732 | 721
Fold rise
  Serotype 1: number analyzed (Participants) | 732 | 720
  Serotype 1 | 7.3 [6.9 to 7.8] | 7.1 [6.7 to 7.6]
  Serotype 3 | 8.5 [7.9 to 9.1] | 9.0 [8.4 to 9.6]
  Serotype 4: number analyzed (Participants) | 731 | 721
  Serotype 4 | 15.4 [14.3 to 16.6] | 14.2 [13.1 to 15.3]
  Serotype 6A: number analyzed (Participants) | 732 | 720
  Serotype 6A | 15.2 [14.3 to 16.2] | 14.5 [13.1 to 15.3]
  Serotype 6B: number analyzed (Participants) | 727 | 718
  Serotype 6B | 18.0 [16.8 to 19.3] | 17.0 [15.8 to 18.2]
  Serotype 7F | 6.0 [5.7 to 6.3] | 6.4 [6.0 to 6.8]
  Serotype 9V: number analyzed (Participants) | 732 | 720
  Serotype 9V | 11.8 [11.1 to 12.6] | 11.2 [10.5 to 11.9]
  Serotype 14 | 5.9 [5.4 to 6.3] | 5.0 [4.6 to 5.3]
  Serotype 5 | 8.9 [8.4 to 9.5] | 8.5 [8.0 to 9.0]
  Serotype 18C | 11.3 [10.6 to 12.0] | 11.4 [10.7 to 12.1]
  Serotype 19A: number analyzed (Participants) | 731 | 721
  Serotype 19A | 25.6 [23.8 to 27.6] | 25.6 [23.6 to 27.7]
  Serotype 19F | 13.1 [12.2 to 14.1] | 12.5 [11.6 to 13.5]
  Serotype 23F | 18.1 [16.8 to 19.5] | 19.2 [17.9 to 20.6]
  Serotype 8: number analyzed (Participants) | 732 | 692
  Serotype 8 | 9.1 [8.5 to 9.8] | 1.3 [1.2 to 1.4]
  Serotype 10A: number analyzed (Participants) | 732 | 718
  Serotype 10A | 8.1 [7.6 to 8.7] | 1.1 [1.0 to 1.1]
  Serotype 11A: number analyzed (Participants) | 732 | 719
  Serotype 11A | 9.8 [9.1 to 10.6] | 1.1 [1.0 to 1.2]
  Serotype 12F: number analyzed (Participants) | 732 | 719
  Serotype 12F | 10.0 [9.4 to 10.6] | 1.0 [1.0 to 1.1]
  Serotype 15B: number analyzed (Participants) | 732 | 719
  Serotype 15B | 8.1 [7.5 to 8.7] | 1.2 [1.2 to 1.3]
  Serotype 22F: number analyzed (Participants) | 732 | 719
  Serotype 22F | 8.4 [7.9 to 9.1] | 1.2 [1.1 to 1.3]
  Serotype 33F: number analyzed (Participants) | 732 | 719
  Serotype 33F | 8.8 [8.2 to 9.4] | 1.1 [1.0 to 1.1]

22. Secondary Outcome: Serotype-specific IgG GMFRs From 1 Month After Dose 3 to 1 Month After Dose 4
Description: GMFR of pneumococcal 20vPnC serotypes included: 1, 3, 4, 5, 6A, 6B, 7F, 8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F and 33F. The GMFR from 1 month after Dose 3 to 1 month after Dose 4 were reported from participants in both Dose 3 and Dose 4 evaluable immunogenicity populations.
Time Frame: from 1 month after Dose 3 to 1 month after Dose 4
Population: Dose 3 and Dose 4 evaluable population: participants aged 42-98 days on Dose 1, received the first 3 doses and 4 doses, had at least 1 valid immunogenicity result 27 to 56 days post Dose 3 or Dose 4. "Number of Participants Analyzed"= maximum number of participants in both Dose 3 and Dose 4 evaluable immuno populations that had a valid IgG concentration at both timepoints. "Number Analyzed"= number of participants with valid IgG concentrations at both timepoints for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 704 | 687
Fold rise
  Serotype 1: number analyzed (Participants) | 704 | 685
  Serotype 1 | 2.0 [1.9 to 2.1] | 1.8 [1.7 to 1.9]
  Serotype 3: number analyzed (Participants) | 704 | 686
  Serotype 3 | 1.6 [1.5 to 1.7] | 1.7 [1.6 to 1.8]
  Serotype 4: number analyzed (Participants) | 703 | 686
  Serotype 4 | 5.1 [4.8 to 5.5] | 4.4 [4.1 to 4.8]
  Serotype 5: number analyzed (Participants) | 704 | 686
  Serotype 5 | 2.9 [2.7 to 3.1] | 2.6 [2.4 to 2.8]
  Serotype 6A: number analyzed (Participants) | 704 | 686
  Serotype 6A | 4.7 [4.4 to 5.0] | 4.3 [4.0 to 4.6]
  Serotype 6B: number analyzed (Participants) | 700 | 685
  Serotype 6B | 6.8 [6.2 to 7.4] | 5.5 [5.0 to 6.0]
  Serotype 7F: number analyzed (Participants) | 704 | 686
  Serotype 7F | 2.3 [2.2 to 2.4] | 2.2 [2.1 to 2.3]
  Serotype 9V: number analyzed (Participants) | 704 | 685
  Serotype 9V | 4.0 [3.7 to 4.3] | 3.4 [3.2 to 3.7]
  Serotype 14: number analyzed (Participants) | 703 | 686
  Serotype 14 | 2.6 [2.4 to 2.9] | 2.2 [2.0 to 2.5]
  Serotype 18C: number analyzed (Participants) | 704 | 686
  Serotype 18C | 2.7 [2.5 to 2.8] | 2.6 [2.5 to 2.8]
  Serotype 19A: number analyzed (Participants) | 703 | 686
  Serotype 19A | 4.9 [4.6 to 5.2] | 4.6 [4.2 to 4.9]
  Serotype 19F: number analyzed (Participants) | 704 | 686
  Serotype 19F | 3.2 [3.0 to 3.4] | 2.9 [2.7 to 3.1]
  Serotype 23F: number analyzed (Participants) | 704 | 686
  Serotype 23F | 4.9 [4.5 to 5.3] | 4.9 [4.5 to 5.3]
  Serotype 8: number analyzed (Participants) | 704 | 659
  Serotype 8 | 2.2 [2.0 to 2.3] | 1.8 [1.6 to 2.0]
  Serotype 10A: number analyzed (Participants) | 704 | 686
  Serotype 10A | 5.3 [4.9 to 5.8] | 1.0 [0.9 to 1.1]
  Serotype 11A | 2.6 [2.4 to 2.8] | 1.1 [1.0 to 1.3]
  Serotype 12F | 3.3 [3.1 to 3.6] | 1.0 [1.0 to 1.1]
  Serotype 15B | 2.8 [2.6 to 3.0] | 1.0 [0.9 to 1.1]
  Serotype 22F | 2.9 [2.7 to 3.1] | 1.0 [0.9 to 1.1]
  Serotype 33F: number analyzed (Participants) | 704 | 686
  Serotype 33F | 6.4 [5.9 to 7.0] | 0.8 [0.8 to 0.9]

23. Secondary Outcome: Percentage of Participants With Alternative Prespecified Hib Antibody Level 1 Month After Dose 3
Description: Antibody concentration to the Hib vaccine antigens were determined on sera collected from a randomly selected subset of participants with sufficient sera volumes. Percentage of participants with alternative prespecified Hib antibody (≥1.0 μg/mL) were reported from Dose 3 evaluable immunogenicity participants.
Time Frame: 1 month after Dose 3
Population: Dose 3 evaluable population: eligible participants aged 42-98 days on Dose 1, received the first 3 doses, had at least 1 valid immunogenicity result within 27 to 56 days post Dose 3, and had no other major protocol deviations. "Number of Participant Analyzed" = Dose 3 evaluable immunogenicity population with valid Hib antibody level. "Number Analyzed" = number of participants with valid Hib antibody level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 124 | 125
percentage of participants | 75.0 [66.4 to 82.3] | 72.0 [63.3 to 79.7]

24. Secondary Outcome: Geometric Mean Ratios (GMRs) of Prespecified Antibody Levels to Specific Concomitant Vaccine Antigen (Measles) 1 Month After Dose 4
Description: Antibody concentrations to concomitant vaccine antigen (measles) were determined on sera collected 1 month after Dose 4 from a randomly selected subset of participants with sufficient sera volumes. GMs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution and were reported from Dose 4 evaluable immunogenicity participants.
Time Frame: 1 month after Dose 4
Population: Dose 4 evaluable immunogenicity population: eligible participants aged 42-98 days on Dose 1, received all 4 doses, have at least 1 valid immunogenicity result within 27 to 56 days after Dose 4, and had no other major protocol deviations as determined by the clinician. "Number of Participants Analyzed"=number of participants in Dose 4 evaluable immunogenicity population with valid antibody concentrations for the specified antigen reported at 1 month after Dose 4.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 234 | 232
AU/mL | 277.74 [243.88 to 316.30] | 215.41 [184.61 to 251.35]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Measles: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - 13vPnC) of the logarithms of the concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR of 20vPnC group to 13vPnC group is greater than 0.5 (2-fold NI margin); Geometric Mean Ratios = 1.29, 95% CI [1.05 to 1.58]

25. Secondary Outcome: GMRs of Prespecified Antibody Levels to Specific Concomitant Vaccine Antigen (Mumps) 1 Month After Dose 4
Description: Antibody concentrations to concomitant vaccine antigen (mumps) were determined on sera collected 1 month after Dose 4 from a randomly selected subset of participants with sufficient sera volumes. GMs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution and were reported from Dose 4 evaluable immunogenicity participants.
Time Frame: 1 month after Dose 4
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 234 | 232
AU/mL | 36.96 [30.82 to 44.33] | 34.19 [28.94 to 40.39]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Mumps: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - 13vPnC) of the logarithms of the concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; Geometric Mean Ratios = 1.08, 95% CI 2-sided [0.85 to 1.38]

26. Secondary Outcome: GMRs of Prespecified Antibody Levels to Specific Concomitant Vaccine Antigens (Rubella) 1 Month After Dose 4
Description: Antibody concentrations to concomitant vaccine antigen (rubella) were determined on sera collected 1 month after Dose 4 from a randomly selected subset of participants with sufficient sera volumes. GMs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution and were reported from Dose 4 evaluable immunogenicity participants.
Time Frame: 1 month after Dose 4
Population: Dose 4 evaluable immunogenicity population: eligible participants aged 42-98 days on Dose 1, received all 4 doses, had at least 1 valid immunogenicity result within 27 to 56 days after Dose 4, and had no other major protocol deviations as determined by the clinician. "Number of Participants Analyzed"= number of participants in Dose 4 evaluable immunogenicity population with valid antibody concentrations for the specified antigen reported at 1 month after Dose 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 234 | 232
IU/mL | 49.63 [43.88 to 56.13] | 40.44 [35.19 to 46.48]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Rubella: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - 13vPnC) of the logarithms of the concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; Geometric Mean Ratios = 1.23, 95% CI 2-sided [1.02 to 1.48]

27. Secondary Outcome: GMRs of Prespecified Antibody Levels to Specific Concomitant Vaccine Antigen (Varicella) 1 Month After Dose 4
Description: Antibody concentrations to concomitant vaccine antigen (varicella) were determined on sera collected 1 month after Dose 4 from a randomly selected subset of participants with sufficient sera volumes. GMs and 2-sided CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs based on the Student's t distribution and were reported from Dose 4 evaluable immunogenicity participants.
Time Frame: 1 month after Dose 4
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 20vPnC | 13vPnC
Number analyzed (Participants) | 231 | 229
mIU/mL | 233.05 [207.25 to 262.06] | 234.78 [208.84 to 263.94]
Statistical Analysis 1: Comparison: 20vPnC vs 13vPnC; Varicella: GMR and 2-Sided CI were calculated by exponentiating the mean difference (20vPnC - 13vPnC) of the logarithms of the concentrations and the corresponding CI (based on the Student's t distribution); Test type: Non-Inferiority — [test comment as in outcome 24, analysis 1]; Geometric Mean Ratios = 0.99, 95% CI 2-sided [0.84 to 1.17]

ADVERSE EVENTS:
Time Frame: Local reactions (LR) and systemic events (SE) [systematic assessment(SA)]:within 7 days after Dose 1, 2, 3, 4; SAEs: from Dose 1 up to 6 months after Dose 4; other AEs [non-systematic assessment (non-SA)]:from Dose 1 up to 1 month after Dose 3 and from Dose 4 up to 1 month after Dose 4
Description: Same events may appear as both an AE and a SAE. However, what are presented are distinct events. An event may be classified as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a SAE and non-SAE during the study
Arm/Group | 20vPnC | 13vPnC
All-Cause Mortality (participants affected / at risk) | 0/1001 | 0/987
Serious Adverse Events (participants affected / at risk) | 45/1001 | 31/987
Other Adverse Events (participants affected / at risk) | 966/1001 | 939/987
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20vPnC (N=1001) | 13vPnC (N=987)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 4 (6) | 4 (4)
Bullous impetigo (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 5 (5)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (2) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 1 (1)
Metapneumovirus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 7 (7) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 5 (5) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2) | 2 (2)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20vPnC (N=1001) | 13vPnC (N=987)
Injection site erythema (REDNESS) (General disorders) | 498 (944) | 492 (986)
Injection site pain (PAIN) (General disorders) | 689 (1634) | 663 (1543)
Injection site swelling (SWELLING) (General disorders) | 353 (635) | 359 (707)
Pyrexia (FEVER) (General disorders) | 322 (550) | 314 (504)
Otitis media (Infections and infestations) | 56 (73) | 50 (65)
Upper respiratory tract infection (Infections and infestations) | 114 (137) | 112 (137)
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 521 (1041) | 492 (1028)
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 823 (2309) | 798 (2268)
Irritability (IRRITABILITY) (Psychiatric disorders) | 894 (3380) | 863 (3301)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04382326/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT04382326/SAP_001.pdf